CLINICAL TRIAL: NCT01406171
Title: A Phase 1, Open-Label, Drug Interaction Study of the Pharmacokinetics of Isavuconazole and Midazolam After Separate and Concomitant Administration to Healthy Adult Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica (Industry)
Responsible Party: Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0023
Record Dates: First submitted 2011-07-06; First posted 2011-08-01 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Pharmacokinetics of Isavuconazole; Pharmacokinetics of Midazolam; Healthy Volunteers
Keywords: Isavuconazole; ASP9766; BAL8557; Midazolam; Healthy volunteers
MeSH Terms: interventions — isavuconazole; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and Midazolam (Experimental): Isavuconazole three times per day (TID) for 2 days followed by once a day (QD) for 9 days. Midazolam single doses on days 1 and 12
  Interventions: Drug: Isavuconazole; Drug: Midazolam

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: ASP9766; BAL8557
Drug: Midazolam — Oral

SUMMARY:
The purpose of this study is to determine the effect of isavuconazole at steady state on the pharmacokinetics of midazolam in healthy adult subjects.

DETAILED DESCRIPTION:
Subjects will check-in on Day -1 and remain confined to the study center until the completion of study procedures on Day 14. Subjects will return to the study center for an outpatient follow-up visit on Day 21. Blood and urine samples will be taken at various times during the study.

Subjects will receive a single dose of oral midazolam syrup on Day 1. On Days 3 and 4, isavuconazole will be dosed orally three times daily (TID). On Days 5 through 13, isavuconazole will be dosed orally once daily (QD). A single dose of oral midazolam syrup will be administered on Day 12.

ELIGIBILITY:
Inclusion Criteria:

* The subject agrees to sexual abstinence, is surgically sterile, is postmenopausal, or is using a medically acceptable method to prevent pregnancy during the study period
* The subject must weigh at least 45 kg and have a body mass index (BMI) of 18-32 kg/m2
* The subject's has a normal 12-lead electrocardiogram (ECG)
* The subject is a non-smoker and has not used tobacco or nicotine products for a minimum of 6 months
* The subject's clinical laboratory test results are within normal limits

Exclusion Criteria:

* The subject has a previous history of any clinically significant gastro-intestinal, neurological, renal, hepatic, pulmonary, metabolic, cardio-vascular, psychiatric, endocrine, hematological disorder or disease, malignancy excluding non-melanoma skin cancer
* The subject has a known or suspected hypersensitivity to midazolam, isavuconazole, or the azole class of compounds
* The subject has a history of consuming more than 14 units of alcoholic beverages per week, has a history of drug or alcohol abuse within the past 2 years, or has a positive screen for alcohol or drugs of abuse/illegal drugs (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to study drug administration, or over-the-counter medication within 1 week prior to study drug administration, with the exception of acetaminophen up to 2g/day
* The subject anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinic admission and throughout the duration of the study
* The subject anticipates an inability to abstain from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to clinic admission and throughout the duration of the study
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission
* The subject has a positive test for hepatitis C antibody or hepatitis B surface antigen or a known history of human immunodeficiency virus
* The subject has been vaccinated within 30 days prior to study drug administration
* The subject has received an experimental agent within 30 days or five half-lives, whichever is longer, prior to study drug administration
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days, or donated plasma within 7 days prior to clinic admission
* The subject has any other condition which precludes the subject's participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic assessment of AUC through the analysis of blood samples | Up to Day 13
Pharmacokinetic assessment of maximum concentration (Cmax) through the analysis of blood samples | Up to Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance Clinical Research, Madison, Wisconsin, United States